CLINICAL TRIAL: NCT02437058
Title: Validition of Scales for the Assessment of Sverity in Acute Decompensated Heart Failure
Brief Title: Validity of Scales to Assess Severity in Acute Heart Failure
Acronym: AHFRS
Status: Completed | Type: Observational
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Collaborators: Hospital Donostia (Other); Hospital de Basurto (Other)
Responsible Party: Principal Investigator, Susana García Gutiérrez, MD,PhD, Hospital Galdakao-Usansolo
Other Study IDs: 2011111045
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: preidictive model

SUMMARY:
The scales measuring the severity of acute decompensate heart failure (ADHF) in emergency departments have not achieved an adequate discriminative ability for decision making. Objectives: 1) Identify baseline variables, and evolutionary variables that may provide a good predictive ability of the model.2) Create and validate clinical predictive rules of mortality during admission/a week after ED visit in those discharged from ED, 30 and 60 days after ED visit as well as identify predicitive factors of short-term readmission (90 days)Design: Prospective cohort study. The sociodemographics and clinical variables will be collected from emergency medical records to identify predictors. Outcome variables and evolution of variables will be collected from hospital medical records / ambulatory during admission and up to 90 days after the episode of ADHF. Baseline predictors and evolutionary variables will be identified through logistic regression models using 60% of the final sample. The models that best fit will be applied in 40% of the sample to assess the predictive validity of this scale.

ELIGIBILITY:
Inclusion Criteria:

* They were diagnosed as heart failure) HF is defined, clinically, as a syndrome in which patients have typical symptoms (e.g.breathlessness, ankle swelling, and fatigue) and signs (e.g. elevated jugular venous pressure, pulmonary crackles, and displaced apex beat) resulting from an abnormality of cardiac structure or function.(8) We included the following presentation of acute heart failure (AHF) at ED: acute decompensated heart failure, hypertensive acute heart failure, pulmonary oedema, cardiogenic shock, and high output failure. (9;10)

Exclusion Criteria:

* Patients whose main diagnosis in the ER is different than acute heart failure and those not wishing to participate in the study or signing the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptoms of acute decompensated heart failure who attended the emergency departments of 3 hospitals belonging to the Basque National Health Service
Sampling Method: Non-Probability Sample
Enrollment: 1854 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Poor evolution | 3 months

SECONDARY OUTCOMES:
readmission | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose María Quintana, PhD, Study Director — Chief of Research unit

REFERENCES:
- [Derived] Garcia-Gutierrez S, Quintana JM, Anton-Ladislao A, Gallardo MS, Pulido E, Rilo I, Zubillaga E, Morillas M, Onaindia JJ, Murga N, Palenzuela R, Ruiz JG; AHFRS Group. Creation and validation of the acute heart failure risk score: AHFRS. Intern Emerg Med. 2017 Dec;12(8):1197-1206. doi: 10.1007/s11739-016-1541-4. Epub 2016 Oct 11. PMID 27730492